CLINICAL TRIAL: NCT05945719
Title: Discrimination and Harassment of Pain Clinic Staff Caused by Patients
Brief Title: Discrimination Harassment of Pain Staff Caused by Patient
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Salem2020 Discrimination By Pt
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Abuse, Sexual; Abuse, Workplace
Keywords: Harassment by patients
MeSH Terms: conditions — Coitus; Occupational Stress | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Adult chronic pain patients who sexually harass pain clinic staff
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral therapy — Behavioral and supportive therapy

SUMMARY:
Chronic pain is associated with mental disorders, and some patients have behavioral issues. Some patients may sexually or racially harass pain clinic staff. Healthcare staff do not usually report sexual or racial harassment perpetrated by patients.

Quantitative and qualitative analysis of prospective electronic and clinic diary data. Evaluation of incidents of sexual and racial harassment of clinic staff; perpetrated by patients. Analysis of causative factors, incident outcome, system factors and lessons learned.

DETAILED DESCRIPTION:
Chronic pain disorder may be associated with mental health disease. Many patients exhibit behavioral problems. Some of the patients may sexually or racially harass the pain clinic staff. Typically, healthcare providers do not report racial or sexual harassment perpetrated by patients.

This is a quantitative analysis of prospective electronic and clinic diary data. It evaluates many incidents of sexual and racial harassment of pain clinic staff; perpetrated by patients. It analyzes the incident causative factors, incident outcomes, system factors and lessons learned. The qualitative information of each incident is presented in a sensitive and careful format.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients

Exclusion Criteria:

* pediatric chronic pain patients

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain patients who are undergoing treatment in a specialist pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who sexually or racially harassed clinic staff | 12 months
  Percentage of patients who sexually or racially harassed clinic staff

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler M, Vincent-Hoper S, Vaupel C, Gregersen S, Schablon A, Nienhaus A. Sexual Harassment by Patients, Clients, and Residents: Investigating Its Prevalence, Frequency and Associations with Impaired Well-Being among Social and Healthcare Workers in Germany. Int J Environ Res Public Health. 2021 May 13;18(10):5198. doi: 10.3390/ijerph18105198. PMID 34068346